CLINICAL TRIAL: NCT05342012
Title: The Effect of Inorganic Nitrate Supplementation on Brown Fat Activation and Quantity in People With Type 2 Diabetes Mellitus
Brief Title: The Effect of Nitrate on Brown Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: University of Portsmouth (Other); Institute of Bioengineering and Bioimaging (IBB) (Other Government); Loughborough University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 306840
Record Dates: First submitted 2022-03-01; First posted 2022-04-22 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Beetroot; Brown Adipose Tissue; Infrared spectrometry; Magnetic Resonance Imaging; Nitrates; Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind randomised control trial. Supplements will be dispensed by a member of the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Beetroot juice then nitrate depleted beetroot juice (Experimental): Participants will be asked to consume 140ml of beetroot juice prior to their first experimental visit. Participants will then be asked to consume 140ml a day for 2 weeks, and finally visit the investigators once more following another 140ml drink.
  Interventions: Dietary Supplement: Concentrated beetroot juice; Dietary Supplement: Nitrate depleted beetroot juice
- Experimental: Nitrate depleted beetroot juice then beetroot juice (Experimental): Participants will be asked to consume 140ml of placebo prior to their first experimental visit. Participants will then be asked to consume 140ml a day for 2 weeks, and finally visit the investigators once more following another 140ml drink.
  Interventions: Dietary Supplement: Concentrated beetroot juice; Dietary Supplement: Nitrate depleted beetroot juice

INTERVENTIONS:
Dietary Supplement: Concentrated beetroot juice — Acute and chronic supplementation of beetroot juice.
Dietary Supplement: Nitrate depleted beetroot juice — (Nitrate depleted beetroot juice

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a metabolic condition characterized by chronic hyperglycemia and progressive insulin resistance, which progressively lead to macro- and microvascular damage. With the number of people with T2DM continuing to rise, this pandemic is expected to reach 700 million people by 2045, such that the costs associated with its clinical management are likely to become unsustainable. Therefore, identifying cost effective alternative interventions is imperative.

Diets rich in fruits and vegetables are well known to have cardiovascular benefits and reduce the risk of getting T2DM. The beneficial effects of vegetables on cardiovascular outcomes are particularly effective in green leafy vegetables and beetroot. This may in part be due to a high concentration of inorganic nitrate, and its beneficial effects on cardiovascular health due to its effect on nitric oxide (NO•). Increased dietary nitrate intake elevates cyclic guanosine monophosphate [(cGMP)]. Importantly, cGMP has also been shown to increase brown fat expression by 'beiging' WAT in mice through an NO• dependent process.

Recent developments in the ability to non-invasively measure BAT activation using magnetic resonance imaging (MRI) and infrared thermography (ITR) has opened the possibility to study the effects of nitrate on BAT activation in man. BAT depots in humans with T2DM have been identified using MRI but not yet with the more easily accessible technique of IRT.

It is hypothesised that nitrate can increase BAT activation and quantity in people with T2DM.

DETAILED DESCRIPTION:
Dietary inorganic nitrate is converted in a reversible, stepwise reaction to nitrite via bacteria on the dorsum of the tongue. Subsequently, small quantities of NO• are produced in the stomach. The remaining nitrite is then absorbed into the circulation where it acts as a storage pool for subsequent NO• production. Production of NO• from nitrite reduction is expedited in hypoxaemia, a phenomenon observed in the vasculature of white adipose tissue (WAT).

WAT is primarily an energy store, whereas brown adipose tissue (BAT) is a metabolically active tissue. BAT is responsible for ~5% of basal metabolic rate and ~15% of total energy expenditure, equating to ~40 g of BAT per day and is used in non-shivering thermogenesis. BAT is used for heat production and is stimulated by cold environments and or diet to cause thermogenesis. To produce heat during cold exposure, uncoupling protein (UCP)-1, an inner mitochondrial protein, is upregulated in BAT ultimately uncoupling the mitochondrial proton gradient, making the cell less energy efficient. Inorganic nitrate supplementation has also been shown to increase UCP-1 expression in BAT.

ELIGIBILITY:
Inclusion Criteria:

* Males or women with Type 2 Diabetes Mellitus

Exclusion Criteria:

* Individuals with a BMI over 30
* Individuals with severe claustrophobia (this would make imaging the BAT less reliable)
* Current smokers (or those that have smoked within 3 months)
* Proton pump inhibitors or phosphodiesterase inhibitor users, as these may affect [cGMP]. Half life of this drug is short. Participants can choose to not use this if they wish to participate.
* Individuals with any other serious medical condition which would interfere with data interpretation or safety will be excluded from participation.
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
MRI Imaging of Supraclavicular BAT | MRI on day 14 (Visit 2) before 60 minutes of cold exposure, following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  High-resolution 3-dimensional T1-weighted imaging will be acquired using repetition time, echo time and field of view.
  All imaging sequences will have anatomical coverage of the neck, supraclavicular region and the apices of the lung.
MRI Imaging of Supraclavicular BAT | MRI on day 14 (Visit 2) following 60 minutes of cold exposure, following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  High-resolution 3-dimensional T1-weighted imaging will be acquired using repetition time, echo time and field of view.
  All imaging sequences will have anatomical coverage of the neck, supraclavicular region and the apices of the lung.
MRI Imaging of Supraclavicular BAT | MRI on day 35 (visit 3) before 60 minutes of cold exposure, following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  High-resolution 3-dimensional T1-weighted imaging will be acquired using repetition time, echo time and field of view.
  All imaging sequences will have anatomical coverage of the neck, supraclavicular region and the apices of the lung.
MRI Imaging of Supraclavicular BAT | MRI on day 35 (visit 3) following 60 minutes of cold exposure, following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  High-resolution 3-dimensional T1-weighted imaging will be acquired using repetition time, echo time and field of view.
  All imaging sequences will have anatomical coverage of the neck, supraclavicular region and the apices of the lung.
A 3D multi-point Dixon sequence will be utilized for the water-fat imaging. | At start of MRI Imaging of Supraclavicular BAT
  A 3D multi-point Dixon sequence will be utilized for the water-fat imaging.
A 3D multi-point Dixon sequence will be utilized for the water-fat imaging. | At end of MRI Imaging of Supraclavicular BAT
  A 3D multi-point Dixon sequence will be utilized for the water-fat imaging.
Pixel wise quantification of fat fraction will be performed from fat and water maps. | At time of MRI Imaging
  Pixel wise quantification of fat fraction will be performed from fat and water maps.

SECONDARY OUTCOMES:
IRT Imaging of Supraclavicular BAT | IRT on day 14 (Visit 2) and day 35 (visit 3), before and after 60 minutes of cold water immersion, following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  Bilaterally, two regions will be analysed for skin temperature from thermal images using infrared cameras: 1) the skin area overlaying BAT in the SCV fossae on the left and right sides, and; 2) the sternal area considered as a control.
Biomarkers - Nitrate | Blood sampling on day 14 (Visit 2) and day 35 (visit 3) following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  Quantified using a Sievers nitric oxide analyser
Biomarkers - Nitrite | Blood sampling on day 14 (Visit 2) and day 35 (visit 3) following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  Quantified using a Sievers nitric oxide analyser
Biomarkers - cGMP | Blood sampling on day 14 (Visit 2) and day 35 (visit 3) following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  Quantified using a Sievers nitric oxide analyser
Biomarkers - Nitrate | Blood sampling on day 14 (Visit 2) and day 35 (visit 3) following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  Quantified using commercially available ELISA assays
Biomarkers - Nitrite | Blood sampling on day 14 (Visit 2) and day 35 (visit 3) following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  Quantified using commercially available ELISA assays
Biomarkers - cGMP | Blood sampling on day 14 (Visit 2) and day 35 (visit 3) following 14-days beetroot/placebo supplementation with 7-day washout between crossover.
  Quantified using commercially available ELISA assays

CONTACTS AND LOCATIONS:
Overall Officials: Rebecc Neal, Study Chair — Senior Lecturer in Exercise Physiology
Locations (4):
- United Kingdom (4):
  - Bournemouth University, Bournemouth, Dorset
  - University of Portsmouth, Portsmouth, Hampshire
  - Southern Health NHS Foundation Trust, Southampton, Hampshire
  - Shore Medical, Poole